CLINICAL TRIAL: NCT04357886
Title: The Comparison of New Coronavirus (COVID-19) Awareness in Individuals of Different Age Groups: Analysis of Turkey
Brief Title: Awareness of COVID-19 in Turkey
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Saliha Gürdal Karakelle, Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: 60350273-605.99-
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: COVID-19; Pandemic; Knowledge and Awareness; Adolescent; Adults
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Because COVID-19 is a new virus, it is believed that awareness assessment will inform and guide what steps should be taken and which groups should be targeted in terms of controlling the pandemic. According to our hypothesis, COVID-19 awareness of individuals in different age groups in the Turkish population also varies. There are controlling pratices based on scientific studies made during the outbreak, but there is no certainty as to how much these measures are known by our society. Based on these, the aim of our study was to investigate and compare the awareness of new Coronavirus (COVID-19) in different age groups across Turkey.

DETAILED DESCRIPTION:
Statistical Analysis: In the statistical analysis of the data obtained at the end of the study, SPSS (Statistical Package for Social Sciences / SPSS 21.0) was analyzed using the statistical program. In the study, arithmetic averages are presented with tables and graphs as mean ± SD (standard deviation) and values indicated by counting in numbers (percent). Demographic information of the participants and their responses to the questionnaire questions were evaluated using descriptive statistical analysis method. In the study, Independent Sample t Test was used in parametric data and ANOVA was used in normal non-parametric data. In all analyzes, p <0,05 was considered statistically significant.

Sampling: Sample size was calculated based on the number of questions asked. Accordingly, the number of questions multiplied by the formula of 60 is the lower limit (42*60=2520). Considering the 20% probability of a drop-out and the fact that participants did not want to volunteer, it was decided to take 3150 people to the study. Consent will be obtained from the participants through a voluntary information form.

ELIGIBILITY:
Inclusion Criteria:

* Having at least primary education
* Being literate in Turkish
* There is a level of cooperation to understand the evaluations
* Agree to participate in the study

Exclusion Criteria:

* Those with audio and visual problems that prevent communication

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: people of diffirent age groups throughout Turkey
Sampling Method: Non-Probability Sample
Enrollment: 2605 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
COVID-19 Awareness Survey | once at baseline of study
  The questionnaire was prepared by the researchers. There are 49 questions in the survey and all of them are multiple choice. The survey assesses the demographic characteristics, awareness and attitudes of the participants towards the COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Ipek Yeldan, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Li H, Liu SM, Yu XH, Tang SL, Tang CK. Coronavirus disease 2019 (COVID-19): current status and future perspectives. Int J Antimicrob Agents. 2020 May;55(5):105951. doi: 10.1016/j.ijantimicag.2020.105951. Epub 2020 Mar 29. PMID 32234466
- See also: access to current data about the COVID-19 in the world — http://who.sprinklr.com
- See also: access to current data about the COVID-19 in Turkey — http://covid19.saglik.gov.tr/